CLINICAL TRIAL: NCT00130455
Title: A 12 Week Multi-Centre, Randomized, Double-Blind, Placebo Controlled Evaluation of the Most Efficacious and Tolerable Dose of Escitalopram in the Treatment of Elderly Patients
Brief Title: Treatment of Depression in the Elderly
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Psychiatric Hospital, Hillerod (Other)
Collaborators: Psychogeriatric Unit, CU Hospital, Frederiksberg (Unknown); Amager Hospital (Other); Psychiatric Center Ballerup (Other); Geriatric Department,Korsør, Vestsjælland (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIL-01
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2007-02-06 (Estimated); Status verified 2007-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
The study is designed to establish the efficacy and tolerability of escitalopram in the treatment of depressive episodes of mild to moderate severity in the elderly.

The study is designed as a mainly naturalistic study including all patients of 65 years of age or above that judged by the clinician would benefit from treatment by an antidepressant medication. The study is designed as a double-blind, randomised placebo controlled study with two groups of active treatment (escitalopram in two doses, 5 or 10 mg daily) in a twelve week period.

ELIGIBILITY:
Inclusion Criteria:

* In- or out-patients of 65 years of age or above fulfilling the International Classification of Diseases-Tenth Edition (ICD-10) diagnosis of depressive single episode (F32.00-32.11. 32.8 or 32.9), depressive recurrent episode (F33.00-33.11, 33.8 or 33.9) or organic depressive episode (F06.32).
* The depressive state should be mild to moderate and reach a score on HAM-D6 of ≥ 7 and ≤ 11
* Patients with dementia can be included provided they have a mini mental state exam (MMSE) score of ≥ 17

Exclusion Criteria:

* Patients with a current depressive episode of a severity reaching a score of ≥ 12 on the HAM-D6-item depression factor. This is to exclude patients with severe or psychotic depression
* Patients with suicidal thoughts or behaviour
* Patients with conditions where treatment with escitalopram is contraindicated: e.g. hypersensitivity to escitalopram or other contents of escitalopram tablets, concomitant treatment with non-selective, irreversible mono-amine-oxidase inhibitors, such as Marplan
* Patients who in the current depressive episode have had a failed trial of treatment with escitalopram
* Co-morbid dementia with a severity corresponding to a score on the MMSE of less than 17 as these patients will often be without the ability to give informed consent
* Patients with sensory defects rendering psychometric assessment impossible, e.g. deafness, blindness, severe aphasia
* Patients who cannot speak Danish well enough to make psychometric assessment possible and meaningful
* Patients with congenital or early acquired intellectual deficits

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 189
Dates: Start 2006-04; Study Completion 2008-01

PRIMARY OUTCOMES:
Remission during the study is defined as a Hamilton 6-item depression subscale (HAM-D6) score less than or equal to 4
Response will be defined as a drop in HAM-D6 score of 50% or more

CONTACTS AND LOCATIONS:
Overall Officials: Alex Koerner, MD, Principal Investigator — Psychiatric hospital, Hilleroed, Denmark
Locations (1):
- Alex Koerner, Hilleroed, Denmark